CLINICAL TRIAL: NCT06350201
Title: Machine Learning-based Classification of Symptom Clusters and Matched Online Cognitive Behavior Intervention for Depression Symptom and Anxiety Symptom
Brief Title: Machine Learning-based Classification of Symptom Clusters and Online CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Mental Health Centre (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY2024.0124.02
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Depression and Anxiety Symptom
Keywords: machine learning approach; CBT; PST; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 weeks Problem-solving therapy (Experimental): Problem-solving therapy imparts problem-solving abilities applicable to participants' daily lives.
  Personalized therapies, including brief behavioral treatment of insomnia, mindfulness, and physical exercise suggestions, were tailored to correspond with patients' specific clusters of sadness and anxiety symptoms.
  Interventions: Behavioral: problem solving therapy
- treatment as usual (Placebo Comparator): Care as usual with the PST-PC learning manual and generic information from the same domains (BBTI, mindfulness, and physical activity) included in the intervention group's daily check-ins
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: problem solving therapy — Problem-solving therapy-based holistic emotion management interventions matched to individual symptoms
  Arms: 8 weeks Problem-solving therapy
Other: control group — Routine psychological care and guidance on mood management
  Arms: treatment as usual

SUMMARY:
To breakthrough the bottleneck identified, we will conduct a cross-sectional study to develop a symptom clustering model for depression and anxiety. A wide range of statistical methods as well as machine learning approaches were explored, and a cohesive hierarchical clustering algorithm will be used. After developing the model, a symptom-matched intervention program based on problem solving therapy will be formulated. We are supposed to examine whether its use for personalizing symptom-matched psychological treatment can lead to improved patient outcomes, compared with usual care. This project is expected to provide a new and precise method for the emotion management, which will provide a standardized intervention pathway combining screening with treatment for the management of depression symptom and anxiety symptom. A preciser intervention matched to individual symptoms may provide important insight in improving patient outcome as well as a standardized mood management pathway targeting to the early detection and intervention for community residents.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 64 years. PHQ-9 ≥10 and/or GAD-7 ≥8 at baseline assessment defined as the threshold for caseness.

Exclusion Criteria:

* People will be excluded if they meet any of the following criteria:

  1. They are receiving psychological therapy during an interview for any mental health issue;
  2. currently acutely suicidal or have attempted suicide in the past 2 months, as indicated by PHQ-9 item 9;
  3. cognitively impaired or diagnosed with bipolar disorder or psychosis or experiencing psychotic symptoms; d) dependent on alcohol or drugs; e) living with an unstable or acute medical illness that would interfere with trial participation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The Patient Health Questionnaire (PHQ-9) | Baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 12, week 20, week 32
GAD-7 | Baseline, week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 12, week 20, week 32

SECONDARY OUTCOMES:
PSQI | Baseline, week 1, week 4, week 6, week 8, week 12, week 20, week 32
WHODAS 2.0 | Baseline, week 1, week 4, week 6, week 8, week 12, week 20, week 32
EQ-5D-5L | Baseline, week 1, week 4, week 6, week 8, week 12, week 20, week 32

OTHER OUTCOMES:
remission rate | week 8, week 12, week 20, week 32
  PHQ-9 < 5 AND/OR GAD-7 < 5
SBQ-R | week -1 pre-screening
  It was utilized to assess suicide ideation for exclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, China

IPD SHARING:
Plan to Share IPD: No